CLINICAL TRIAL: NCT05076669
Title: Quality of Life Impact After Enhanced Follow-up of Ostomy Patients by a Home Healthcare Nursing Service Employing Stomal Therapy Nurse Consultants Compared to Conventional Care
Brief Title: Quality of Life Impact After Enhanced Follow-up of Ostomy Patients
Acronym: StomaCare
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: FSK (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSK-001; NCT05061927 (obsolete NCT alias)
Record Dates: First submitted 2021-09-21; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Stoma Ileostomy; Stoma Colostomy; Quality of Life
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Open-label, randomised, comparative, controlled, national and multi-centre study with minimal risks and constraints to routine care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The control group will receive the routine care prescribed by the sites and will be provided with ostomy equipment by FSK.
  Interventions: Other: standard of care
- interventional group (Experimental): The interventional group will benefit from delivery and enhanced follow-up by the FSK HHN provided, in particular, by stomal therapy nurse consultants and patient-relation experts during in-person or remote appointments in addition to the routine care delivered and prescribed by the sites.
  Interventions: Other: stoma follow-up

INTERVENTIONS:
Other: stoma follow-up — delivery and enhanced follow-up by the FSK HHN provided, in particular, by stomal therapy nurse consultants and patient-relation experts during in-person or remote appointments in addition to the routine care delivered and prescribed by the sites
  Arms: interventional group
Other: standard of care — routine management of stoma
  Arms: Control

SUMMARY:
In this context, FSK would like to implement a clinical study to assess the added value on the health-related QoL from the enhanced follow-up of ostomy patients by a HHN including stomal therapists.

The interventional group will benefit from delivery and enhanced follow-up by the FSK HHN provided, in particular, by stomal therapy nurse consultants and patient-relation experts during in-person or remote appointments in addition to the routine care delivered and prescribed by the sites.

The control group will receive the routine care prescribed by the sites and will be provided with ostomy equipment by FSK.

DETAILED DESCRIPTION:
France currently has about 80,000 ostomy patients. Stoma placement exposes patients to many surgical or peristomal skin complications which could impair the quality of life of the ostomy patient.

The management of ostomy patients varies from institution to institution and according to how the patient's medical equipment is supplied as well as whether or not specialised personnel are available.

In the last decade, the market for stoma therapy in France has evolved, with a significant increase in the delivery of equipment by HHNs, meeting a need for patient follow-up and accompaniment.

This increased preference of HHNs to use specialist nurses seems to be explained by the added benefits. Early international studies have demonstrated the impact of an enterostomal therapy nurse follow-up on the improvement of ostomy patient's quality of life (QoL) relative to their health.

However, none of the studies available today on follow-ups performed by an enterostomal therapist included the French population. Furthermore, the studies show methodological gaps, a limited time span and are based on strong hypotheses.

In this context, FSK would like to implement a clinical study to assess the added value on the health-related QoL from the enhanced follow-up of ostomy patients by a HHN including stomal therapists.

The interventional group will benefit from delivery and enhanced follow-up by the FSK HHN provided, in particular, by stomal therapy nurse consultants and patient-relation experts during in-person or remote appointments in addition to the routine care delivered and prescribed by the sites.

The control group will receive the routine care prescribed by the sites and will be provided with ostomy equipment by FSK.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years
* Patients with a stoma placed less than 10 days ago
* Patients who had a stoma during their current hospitalisation
* Patients informed verbally and in writing via the information sheet and who signed the informed consent form.

Exclusion Criteria:

* Patients in palliative care
* Patients participating in another clinical study interested in the management of ostomy patients
* Patients not enrolled in a social security system or with the CMU (Couverture maladie universelle [Universal Health Coverage])
* Patients under judicial protection or under guardianship
* Patients deprived of freedom (in prison and psychiatric patients being treated without consent)
* Patients with difficulties understanding or reading French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 3 months
  score from the Stoma-QOL specific questionnaire (min: 0- max: 100), analysis of the mean

SECONDARY OUTCOMES:
Satisfaction of patient | 3 and 6 months
  scale 0-100
Quality of life | 1, 2, 3 and 6 months
  Stoma-QOL questionnaire, (min: 0- max: 100), analysis of the mean
Quality of life | 1, 2, 3 and 6 months
  EQ-5D-5L questionnaire (min: 0- max: 1), analysis of the mean
Cost | 3 and 6 months
  • Calculation of resource use at 3 and 6 months per expenditure item (use of services, drug use, medical device and home healthcare service use, MCO (Médecine chirurgie obstétrique [Obstetric surgery]) hospitalisations and SSR (Soins de suite et de réadaptation [Follow-up care and rehabilitation]) hospitalisations) for each group.
Morbidity | 3 and 6 months
  readmission rate

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie H Lefevre, MD, PhD, Principal Investigator — Sorbonne University
Locations (10):
- France (10):
  - Hopital Bicètre, Le Kremlin-Bicêtre
  - Hopital Lyon-Sud, Lyon
  - Hopital SAint Louis, Paris
  - Hopital Saint-Louis, Paris
  - Hopital Saint-Antoine, Paris
  - Hopital de la Pitié-Salpétrière, Paris
  - Hopital HEGP, Paris
  - ESPIC FOCH - Digestige Unit, Suresnes
  - ESPIC Foch - Urology Unit, Suresnes
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Becker A, Schulten-Oberborsch G, Beck U, Vestweber KH. Stoma care nurses: good value for money? World J Surg. 1999 Jul;23(7):638-42; discussion 642-3. doi: 10.1007/pl00012361. PMID 10390579
- [Result] Persson E, Berndtsson I, Carlsson E, Hallen AM, Lindholm E. Stoma-related complications and stoma size - a 2-year follow up. Colorectal Dis. 2010 Oct;12(10):971-6. doi: 10.1111/j.1463-1318.2009.01941.x. PMID 19519689
- [Result] Neil N, Inglese G, Manson A, Townshend A. A Cost-Utility Model of Care for Peristomal Skin Complications. J Wound Ostomy Continence Nurs. 2016 Jan-Feb;43(1):62-8. doi: 10.1097/WON.0000000000000194. PMID 26633166
- [Result] Marquis P, Marrel A, Jambon B. Quality of life in patients with stomas: the Montreux Study. Ostomy Wound Manage. 2003 Feb;49(2):48-55. PMID 12598701
- [Result] Danielsen AK, Rosenberg J. Health related quality of life may increase when patients with a stoma attend patient education--a case-control study. PLoS One. 2014 Mar 7;9(3):e90354. doi: 10.1371/journal.pone.0090354. eCollection 2014. PMID 24609004
- See also: Website of FSK — http://fsk.fr